CLINICAL TRIAL: NCT01464229
Title: A Placebo-Controlled Crossover Study of Iloperidone Augmentation of SSRIs for Residual Anger and Irritability in Major Depressive Disorder
Brief Title: Iloperidone Augmentation of SSRIs for Patients With Major Depressive Disorder With Residual Anger and Irritability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maurizio Fava, MD (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Maurizio Fava, MD, Executive Vice Chair, Department of Psychiatry, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P002043
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — iloperidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iloperidone addition to SSRI antidepressant (Experimental)
  Interventions: Drug: Iloperidone
- Placebo addition to standard SSRI antidepressant (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iloperidone — Iloperidone 1-8 mg for 4 weeks
  Arms: Iloperidone addition to SSRI antidepressant
Drug: Placebo — Placebo
  Arms: Placebo addition to standard SSRI antidepressant

SUMMARY:
Iloperidone is an atypical antipsychotic drug, FDA-approved for the acute treatment of schizophrenia in adults in 2009 (Marino et al., 2010); moreover, some of its pharmacological features seem to be very promising in treating symptoms like anger and anxiety (Fava et al., 1997; Wang et al., 2010). The investigators therefore feel that an adequately sized, well powered, double-blind, placebo-controlled, randomized, cross-over study of iloperidone augmentation of SSRIs among MDD outpatients in partial remission with residual anger and irritability is warranted at this point to evaluate its efficacy, safety and tolerability on residual anger, irritability and depressive symptoms.

Main hypothesis: Adults with MDD in partial remission, who are experiencing residual symptoms of anger and irritability, assigned to treatment with iloperidone will demonstrate a significantly greater reduction in the total score of the Anger/Hostility Scale of the Symptom Questionnaire from baseline to endpoint than those assigned to placebo using the cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Men or women ages 18-65 years old.
* Current Major Depressive Episode in partial remission based on the Structured Clinical Interview for DSM IV-Axis I Disorders (SCID I/P) and a HAM-D-17 score between 9 and 15.
* Current treatment with a selective serotonin reuptake inhibitor (SSRI) other than paroxetine or fluoxetine for at least three months, at a stable dose for the past 4 weeks, and more than 50% but less than 75% improvement on the current antidepressant, as determined by the MGH Antidepressant Treatment Response Questionnaire (ATRQ).
* Score > 8 on the Anger/Hostility Scale of the Symptom Questionnaire both at screen and baseline.

Exclusion Criteria:

* The following DSM-IV diagnoses: 1) organic mental disorders; 2) substance use disorders, including alcohol, active within the last 3 months; 3) schizophrenia; 4) delusional disorder; 5) psychotic disorders not elsewhere classified; 6) bipolar disorder; and 9) antisocial personality disorder; 10) dementia.
* Current, serious suicidal or homicidal risk.
* Pregnancy or breast-feeding.
* Serious, unstable medical illness including cardiovascular, kidney, liver, neurological and endocrine disorders.
* Congenital long QT syndrome or a QTc > 450 ms.
* History of cardiac arrhythmias.
* Electroconvulsive therapy (ECT) within the 6 months preceding baseline.
* Concomitant use of buspirone, fluoxetine, paroxetine, any psychostimulant, modafinil, other antipsychotic drugs, or anticonvulsants (although stable doses of benzodiazepines and hypnotics are allowed) (see Concomitant Therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Ionescu DF, Fava M, Kim DJ, Baer L, Shelton RC, Cusin C. A placebo-controlled crossover study of iloperidone augmentation for residual anger and irritability in major depressive disorder. Ther Adv Psychopharmacol. 2016 Feb;6(1):4-12. doi: 10.1177/2045125315618621. PMID 26913173
- See also: Massachusetts General Hospital Depression Clinical and Research Program Website — http://www.massgeneral.org/psychiatry/services/treatmentprograms.aspx?id=1156

RESULTS

PARTICIPANT FLOW:
Groups:
- Iloperidone, Then Placebo: Iloperidone (1-8 mg) for 4 weeks, then placebo for 4 weeks; in addition to standard SSRI antidepressant
- Placebo, Then Iloperidone: Placebo: Placebo for 4 weeks, then iloperidone for 4 weeks; in addition to standard SSRI antidepressant
Period: Overall Study
Arm/Group | Iloperidone, Then Placebo | Placebo, Then Iloperidone
Started | 10 | 10
Completed | 5 | 8
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Iloperidone, Then Placebo: Iloperidone: Iloperidone 1-8 mg for 4 weeks then placebo for 4 weeks, in addition to SSRI antidepressant
- Placebo, Then Iloperidone: Placebo: Placebo for 4 weeks then iloperidone for 4 weeks; addition to standard SSRI antidepressant
- Total: Total of all reporting groups
Arm/Group | Iloperidone, Then Placebo | Placebo, Then Iloperidone | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: 20 patients randomized into the study.
  Participants
    Females: number analyzed (Participants) | 6 | 8 | 14
    Females | 6 | 8 | 14
    Males: number analyzed (Participants) | 4 | 2 | 6
    Males | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: SQ Anger/Hostility Scale
Description: Of the 20 patients randomized, data was analyzed for 13 completers. Symptom Questionnaire (SQ) Anger/Hostility Scale; this is a 23-item subscale of the 92-item Symptom Questionnaire.
  This score ranges from 0 to 23; higher values represent higher anger and hostility.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: Score on Anger/Hostility Scale
Groups:
- Iloperidone, Then Placebo: Iloperidone: Iloperidone 1-8 mg for 4 weeks then placebo for 4 weeks; addition to SSRI antidepressant
Arm/Group | Iloperidone, Then Placebo | Placebo, Then Iloperidone
Number analyzed (Participants) | 5 | 8
Score on Anger/Hostility Scale
  Iloperidone | 4.8 (4.3) | 8 (6.2)
  Placebo | 6.7 (5.8) | 7.5 (7.2)

ADVERSE EVENTS:
Arm/Group | Iloperidone | Placebo
Serious Adverse Events (participants affected / at risk) | 2/13 | 0/13
Other Adverse Events (participants affected / at risk) | 13/13 | 5/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iloperidone (N=13) | Placebo (N=13)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Increased Irritability (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloperidone (N=13) | Placebo (N=13)
Dry Mouth (Skin and subcutaneous tissue disorders) | 6 | 1
Somnolence (Nervous system disorders) | 2 | 2
Headaches (Nervous system disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Cramping (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No